CLINICAL TRIAL: NCT01665508
Title: Nebivolol for the Relief of Microvascular Angina in Women
Brief Title: Study to Evaluate Effect of Nebivolol on Angina in Women With Microvascular Disease
Acronym: NIRVANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Nandita Scott, Co-Director Corrigan Women's Heart Health Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYS-IT-75
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2016-12

CONDITIONS: Microvascular Angina
Keywords: angina; cardiopulmonary testing; metabolomics; nebivolol
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nebivolol (Experimental): Testing will be performed at baseline (SAQ questionnaire, cardiopulmonary testing, resource utilization, metabolomics and vascular testing). This will be repeated on the same group of patients after 3 months of nebivolol treatment.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Patient to start nebivolol and have repeat testing in 3 months
  Other Names: Bystolic

SUMMARY:
Women have less significant blockages of coronary arteries, however have greater symptoms and worse outcomes compared to their age-matched male counterparts. This paradox has led to the recognition and importance of the microvasculature ( small vessels) as a contributor to symptoms and outcomes. Nebivolol has unique antioxidant properties and dilates blood vessels and it is therefore proposed that treatment with nebivolol will reduce angina (chest symptoms) in women with microvascular disease as well as improve exercise capacity, reduce resource utilization and improve other measures of artery function.

DETAILED DESCRIPTION:
Though women have less obstructive coronary artery disease (CAD) they continue to have a greater burden of symptoms, more myocardial ischemia, and a higher rate of adverse outcomes than their age-matched male counterparts. This ostensible paradox has led to the recognition of a distinct pathophysiology of ischemic heart disease, in part related to microvascular dysfunction, and abnormal coronary reactivity. The term primary microvascular angina, (MVA) is used to describe a syndrome among patients who have symptoms suggestive of cardiac ischemia, evidence of electrocardiographic abnormalities, abnormalities on stress imaging or a history of ACS, but no evidence of obstructive epicardial coronary disease. In this population, microvascular angina causes significant morbidity and in some may contribute to increased mortality.

The treatment of microvascular disease remains empirical due to lack of data regarding symptom alleviation, as well as ultimate mortality reduction. Women with ischemic heart disease and microvascular angina continue to report more frequent angina and worse quality of life. They frequently seek medical attention for the evaluation of cardiovascular symptoms including chest pain and shortness of breath. Consequently, these women incur greater healthcare costs, with more office visits, hospitalizations, and myocardial infarctions. In fact, more than one half of women without obstructive coronary disease continue to have ischemic symptoms that lead to further consumption of CAD resources, most often because of diagnostic uncertainty.

In the absence of robust outcomes data to drive the care of these women with microvascular ischemia, various approaches are taken, in addition to the fundamental management of baseline risk factors. Some physicians treat these women as they would treat patients with known obstructive CAD, while some, in the setting of "open" coronary arteries and persistent chest pain, opt for reassurance. Nevertheless, given that these women with microvascular ischemia continue to have higher morbidity and mortality, as well as increased resource consumption, there is a widely recognized need for effective therapeutic agents to reduce symptoms, improve quality of life, decrease resource consumption, and ultimately reduce mortality.

Nebivolol, due to its unique antioxidant and vasodilator properties, via its effect on NO bioactivity, and subsequent effects on the endothelium may be a potentially ideal therapeutic agent for the treatment of microvascular angina among women. For example, one previous study showed that nebivolol improved exercise parameters, as well as endothelial function, more effectively than other beta blockade with metoprolol, among patients with persistent angina and non-obstructive coronary disease.

Cardiopulmonary exercise testing is an ideal diagnostic test in this study as it will provide unique information on how microvascular ischemia influences functional capacity as measured through sensitive gas exchange parameters. Because it is known that a distinct pathophysiology contributes to microvascular angina among this subset of women, these parameters provided by CPET may provide essential information regarding the mechanism of symptom mitigation should nebivolol confer therapeutic value.

Furthermore, because exercise tolerance is often significantly impaired, objective measures of gas exchange that reflect submaximum and maximum fitness among these women will be useful both at baseline and on nebivolol.

Peripheral arterial tone and pulse wave analysis will also be performed. PAT signal technology provides a widely validated measurement of endothelium-mediated changes in vascular tone, using non-invasive bio-sensors on the fingertips that are elicited by creating a down-stream hyperemic response. This parameter correlates well with endothelial dysfunction in coronary arteries. We will perform endothelial function testing at baseline and after 3 months.

Metabolomics is an emerging field that offers the possibility of using the body's metabolites to both phenotype a disease as well as track its response to isolated perturbations, such as administration of a drug. In this study we will utilize metabolomics to define signatures of microvascular ischemia as well as nebivolol-mediated changes in metabolic profiles. Baseline metabolic profiling, as well as metabolic profiling after 3 months of nebivolol treatment will be performed in this study.

This type of assessment is an ideal complement to the clinical parameters delineated above as it combines targeted mass spectrometry to measures small molecules related to nitric oxide metabolism (ie: arginine, arginosuccinate, citrulline, ornithine, cGMP, ADMA) as well as more unbiased screening of metabolites that are not known to be associated with either nebivolol exposure or microvascular angina.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 40-80
* with evidence of coronary microvascular dysfunction as determined by the presence of rest and or exertional chest tightness and a history of either an elevated troponin level or positive stress test ( EKG criteria or imaging) , as well as non-obstructive coronary artery disease (<50% epicardial obstruction) by either diagnostic catheterization with coronary angiography or CT angiography.

Exclusion Criteria:

* Women who cannot tolerate a beta blocker.
* Women receiving Hormone Replacement Therapy
* Women of child-bearing age who are not on a birth-control method.
* Women with inability to exercise.
* Women with left ventricular systolic dysfunction (LVEF less than 40%)
* Women who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
* Women with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
* Women who are unable to speak, read, and understand English and are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.
* Women with any contraindications to beta blocker therapy
* Women with myocardial bridging
* Women with Prinzmetal's angina

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nandita S Scott, MD, Principal Investigator — Massachusetts General Hospital; Malissa J Wood, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol
Started | 12
Completed | 7
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nebivolol
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Seattle Angina Questionnaire Score
Description: Seattle Angina Questionnaire (SAQ):
  The SAQ is a 5 part survey that is widely used and well validated tool to assess angina stability and angina frequency among patients with coronary artery disease.
  The SAQ is a validated, self-administered 19-item questionnaire with 5 different dimensions of health status in patients with CAD including: angina frequency, angina stability, disease-specific quality of life, physical limitations and treatment satisfaction. Each SAQ domain score ranges from 0-100, with higher scores indicating a better health status.
Time Frame: 3 months
Population: 7 patients complete baseline and followup data reported below is anginal stability
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nebivolol: Testing will be performed at baseline (SAQ questionnaire, cardiopulmonary testing, resource utilization, metabolomics and vascular testing). This will be repeated on the same group of patients after 3 months of nebivolol treatment.
  Nebivolol: Patient to start nebivolol and have repeat testing in 3 months
  There was a significant improvement in angina stability (p=0.034) post treatment compared to baseline. The other parameter of the SAQ were not statistically different ( physical limitation, angina frequency, treatment satisfaction and quality of life)
- Baseline: results prior to nebivolol start
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
units on a scale
  anginal stability | 83.3 (25.8) | 29.2 (18.8)
  phyisical limitation | 74.1 (18.0) | 67.6 (21.1)
  anginal frequency | 80.0 (20.0) | 70.0 (15.5)
  treatment satisfaction | 81.3 (18.5) | 84.4 (13.0)
  qualify of life | 62.5 (33.6) | 51.4 (23.2)

2. Secondary Outcome: Peak VO2 Measured by Cardiopulmonary Exercise Testing
Description: Assessment of exercise capacity (peak VO2) as determined by CPET
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ml/beat
Groups:
- Baseline: results off nebivolol
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
ml/beat | 13.1 (2.3) | 11.0 (2.5)

3. Secondary Outcome: Resource Utilization Questionnaire
Description: Resource utilization as determined by patient phone calls, office visits, emergency room visits, and number of hospitalizations, as well an index cost for any hospitalizations
Time Frame: 3 months
Population: data was not collected
Groups:
- Nebivolol: Testing will be performed at baseline (SAQ questionnaire, cardiopulmonary testing, resource utilization, metabolomics and vascular testing). This will be repeated on the same group of patients after 3 months of nebivolol treatment.
  Nebivolol: Patient to start nebivolol and have repeat testing in 3 months
  this data was incomplete and not useful for analysis
Arm/Group | Nebivolol
Number analyzed (Participants) | 0

4. Secondary Outcome: SF36
Description: The SF-36v2 is a commonly used instrument to assess HRQoL8. The questionnaire evaluates 8 HRQoL domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The physical component score is a composite of the SF-36v2 physical health domains (physical functioning, role-physical, bodily pain and general health) and the mental component score a composite of the mental health domains (vitality, social functioning, role-emotional and mental health). Each HRQoL domain score ranges from 0 to 100, with higher scores corresponding to a better health status. The SF-36v2 domain scores were calculated using the QualityMetric Health Outcomes Scoring Software version 4.5.
Time Frame: baseline and 12 week follow-up
Population: physical functioning reported below
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
units on a scale
  physical functioning | 75.0 (13.8) | 67.9 (10.8)
  role-physical | 85.4 (12.9) | 82.3 (16)
  bodily pain | 75.2 (19.9) | 78.7 (22.8)
  general health | 75 (12.6) | 72.8 (11.1)
  vitality | 67.7 (14.5) | 63.5 (15)
  social functioning | 91.7 (10.2) | 91.7 (15.1)
  role-emotional | 90.3 (15.3) | 97.2 (16.8)
  mental health | 81.7 (6.1) | 81.7 (9.3)
  physical component | 50.3 (4.9) | 48.4 (6.3)
  mental component | 55.3 (5) | 56.7 (3.6)
Statistical Analysis 1: Comparison: Nebivolol; Continuous variables were reported as the mean ± (SD) and categorical data presented as frequency and percentage of the sample. Comparisons between baseline and post-treatment SAQ scores, SF-36v2 scores, and CPET variables were performed using a paired t-test for normally distributed variables or a Wilcoxon signed-rank test for non-normally distributed variables. Normality was defined by the Shapiro-Wilk test. For categorical variables, data were compared using a chi-squared test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Exercise Duration
Description: Assessment of exercise duration as determined by CPET
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Baseline: results without nebivolol
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
minutes | 11.9 (1.1) | 11.8 (1.9)

6. Secondary Outcome: Peak Heart Rate as Measured by Cardiopulmonary Exercise Testing
Description: Assessment of peak heart rate as determined by CPET
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
beats per minute | 119 (11) | 145 (17)

7. Secondary Outcome: Peak O2 Pulse
Description: peak O2 pulse as measured by cardiopulmonary exercise testing
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | Nebivolol | Baseline
Number analyzed (Participants) | 7 | 7
ml/beat | 13.1 (2.3) | 11 (2.5)

ADVERSE EVENTS:
Arm/Group | Nebivolol
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No